CLINICAL TRIAL: NCT04073407
Title: A Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Physiological Effects on Liver Structure and Function of an Amino Acid Food Product, AXA1957, in Adolescent Subjects With Fatty Liver
Brief Title: Study of the Safety and Tolerability of AXA1957 in Adolescent Subjects With Non-Alcoholic Fatty Liver Disease (NAFLD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor has determined that information it would have collected would not inform future development of a therapy with AXA 1957 for NAFLD
Sponsor: Axcella Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AXA1957-002
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Results first posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-08

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AXA1957 (Active Comparator): AXA1957 20.4g
  Interventions: Dietary Supplement: AXA1957
- Placebo (Placebo Comparator): Placebo 24g
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AXA1957 — Amino acids, food study
  Arms: AXA1957
Dietary Supplement: Placebo — placebo
  Arms: Placebo

SUMMARY:
This is a randomized, single blind study to determine whether AXA1957, a novel composition of amino acids, is safe and well tolerated. Subjects will be adolescents with non-alcoholic fatty liver disease (NAFLD), and it will also examine liver biology using blood tests and magnetic resonance imaging (MRI).

ELIGIBILITY:
Key Inclusion Criteria:

* Willing to participate in the study and provide written informed consent.
* Male and female adolescent subjects aged 12 to 17 years
* Subjects must not have participated in any diet/lifestyle intervention or observational studies, or engaged in any body weight altering regimens that resulted in body weight fluctuations (i.e. body weight loss or gain by 5%) in the preceding 30 days prior to Screening.
* Non alcoholic fatty liver disease
* Diabetes or prediabetes
* A screening MRI consistent with liver inflammation and fibrosis

Key Exclusion Criteria:

* Current or history of significant alcohol consumption
* History or presence of liver disease (other than NAFLD/NASH)
* History or presence of cirrhosis and/or history or presence of hepatic decompensation
* Any diabetes other than Type 2
* Other poorly controlled medical condition (for example, uncontrolled hypertension with a systolic blood pressure > 100 mmHg)
* Known sensitivity and/or history of clinically significant food intolerance/allergies to proteins (including whey, soy, casein, amino acids, etc.),
* Unable or unwilling to adhere to contraception requirements
* Any contraindications to a MRI scan
* Any other condition that, in the opinion of the Investigator, renders the subject at risk for compliance, compromises the well-being of the subject, or hinders study completion

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2019-07-27 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saul Faust, MBBS MRCPCH PhD, Principal Investigator — University of Southampton
Locations (4):
- United Kingdom (4):
  - Royal London Children's Hospital, London
  - King's College Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Univeristy of Southhampton, Southampton

RESULTS

PARTICIPANT FLOW:
Period: Part 1
Arm/Group | AXA1957 | Placebo
Started | 6 | 3
Completed | 1 | 2
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Subjects discontinued in response to restrictions on the study due to impact of COVID-19 pandemic | 4 | 1
Period: Part 2
Arm/Group | AXA1957 | Placebo
Started | 0 (Following Part 1, all subjects (including those randomly assigned to the placebo arm in Part 1) were given the option to continue in Part 2 to receive the study food product twice daily for an additional 12 weeks. If the subject chose to not take part in Part 2, the subject underwent a safety follow-up visit approximately 2 weeks after Week13 (Visit 6).) | 1 (Following Part 1, all subjects (including those randomly assigned to the placebo arm in Part 1) were given the option to continue in Part 2 to receive the study food product twice daily for an additional 12 weeks. If the subject chose to not take part in Part 2, the subject underwent a safety follow-up visit approximately 2 weeks after Week13 (Visit 6).)
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | AXA1957 | Placebo | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 3 | 9
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (1.38) | 13.7 (1.15) | 13.6 (1.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs).
Description: Study food product emergent adverse events (AEs). Subjects reporting >or equal to 1 study food product-emergent AE.
Time Frame: AEs Baseline to week 13 - Part 1
Population: Safety analysis for Part 1 Baseline to week 13
Measure: Count of Participants; unit: Participants
Arm/Group | AXA1957 | Placebo
Number analyzed (Participants) | 6 | 3
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: From the time of informed consent up to first administration of study product on Day 1, any untoward medical occurrence considered related to study procedures will be recorded as an AE. Adverse events that occur from the first administration of study product on Day 1 through Week 13 (Part 1) and through Week 27 / Follow-up (Part 2 / Optional) will be considered treatment-emergent AEs.
Arm/Group | AXA1957 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 2/6 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXA1957 (N=6) | Placebo (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT04073407/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT04073407/SAP_001.pdf